CLINICAL TRIAL: NCT05104619
Title: Prospective Analysis of Tumor Tissues From the Oral Cavity by SpiderMassTM Spectroscopy
Brief Title: Spectroscopic Analysis of Tongue Tumor Samples.
Acronym: SpecTum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Université de Lille (Other)
Responsible Party: Sponsor
Other Study IDs: s PI2020_843_0156
Record Dates: First submitted 2021-10-12; First posted 2021-11-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Mass Spectroscopy; Molecular Profile; Surgical Margins; Squamous Cell Carcinoma; Oral Cavity; Tongue
Keywords: mass spectroscopy; molecular profile; surgical margins; squamous cell carcinoma; oral cavity; tongue
MeSH Terms: conditions — Margins of Excision; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue samples will be taken from the tumor and the non-tumor areas. Surgical specimens will be taken in a fresh state immediately after surgery, by an anatomopathologist and a pathological anatomy technician. The sample will be analyzed under standard conditions. Two sites will be selected macroscopically (including a tumor area, a dysplasia area, and a non-tumor area).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tumor samples: (SCC of the tongue)
  Interventions: Procedure: tongue surgery
- healthy tissues
  Interventions: Procedure: tongue surgery

INTERVENTIONS:
Procedure: tongue surgery — In squamous cell carcinoma of the tongue, complete surgical resection of the tumor

SUMMARY:
In squamous cell carcinoma of the tongue, complete surgical resection of the tumor generally represents the primary treatment strategy. Among factors determining the disease prognostic, the surgical margins status is essential for the continued management of the patient, with or without complementary therapies. Generally, surgical margins are defined using visual and tactile elements. Unfortunately, in 15 to 30 percent of cases, they are defined as positive after histopathological examination, on average 5 to 7 days post-surgery.

Techniques have recently been developed to analyze the cancerous and non-cancerous nature of tissues, using the spectral properties of tumor cells. SpiderMass™ is an instrument equipped with a probe for tissue micro-sampling and real-time molecular profile analysis. It is thus ultimately a tool for anatomopathological decision support, for diagnosis and prognosis of the disease. Used in the operating room, SpiderMass™ could also become an innovative surgical tool to precisely define cancerous areas in situ and the margins status in intraoperative conditions.

Based on the principle of artificial intelligence, the SpiderMass™ machine must initially learn to recognize pathological tissues versus healthy. This project aims to accomplish this first phase of machine learning for squamous cell carcinoma of the tongue.

ELIGIBILITY:
Inclusion Criteria:

* age : 18 years and older
* squamous cell carcinoma of the tongue
* surgical resection as first-line treatment
* tumor classification T1 to T4.

Exclusion Criteria:

* metastatic disease
* neoadjuvant therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the Maxillofacial Surgery Department of the CHU Amiens-Picardie for a squamous cell carcinoma of the tongue and for whom the first-line treatment is surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Tumor cells detection in tongue tumor with SpiderMass technique | 1 year
  Tumor cells detection in tongue tumor with SpiderMass technique

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No